CLINICAL TRIAL: NCT03150563
Title: Effects of Different Intensities of Passive Static Stretching on Flexibility, Neuromuscular and Functional Performance in Soccer Athletes: A Blinded, Randomized Controlled Trial.
Brief Title: Differents Intensities of Passive Stretching on ROM, Neuromuscular and Performance in Soccer Players: A Blinded RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Wouber Hérickson de Brito Vieira, Clinical Professor, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.883.129
Record Dates: First submitted 2017-05-06; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Contracture of Muscle, Thigh; Muscle Rigidity; Strain of Hamstring Muscle (Disorder)
Keywords: Stretching; Stretching sensation; Isokinetic dynamometry; Stretching load.
MeSH Terms: conditions — Contracture; Muscle Rigidity

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The randomization process of the sample will be carried out through the electronic website http://www.randomization.com, carried out by a subject external to the experimental and evaluation procedures. With this data, the site will generate a specific coding for each group and will randomly distribute the subjects into four groups: Control Group (GC), Experiment Group 1 (GE1), Experiment Group (GE2) and Experiment Group 3 (GE3).
  The distribution will be kept in an opaque and sealed envelope, being revealed only to P2 only at the time of intervention. The P1, who will carry out the measurements, will not know to which group the individual belongs. To maintain the "blinding" procedure of the study, each individual at the time of intervention will spend 10 minutes in the intervention room (being 4 minutes for preparation and 6 minutes for intervention) and each group will have a corresponding color for the convenience of P2 White, blue, green and yellow).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (No Intervention): The subjects of the CG will receive the same orientations of the other groups in relation to the importance of the routines of stretching activities, but during the study period, they will not be able to perform stretches during their day to day life.
- Experimental Group 1 (Experimental): The experimental group 1 will have the sensation of "SENSATION SENSING WITHOUT DESCONFORT" as an intensity for the application of the passive stretch protocol.
  Interventions: Other: Passive static stretch
- Experimental Group 2 (Experimental): The GE2 will have the feeling of "MAXIMUM DISORDER WITHOUT PAIN" as the as an intensity for the application of the passive stretch protocol.
  Interventions: Other: Passive static stretch
- Experimental Group 3 (Experimental): GE3 will have the sensation of "MAXIMUM TOLERABLE PAIN" as the as an intensity for the application of the passive stretch protocol.
  Interventions: Other: Passive static stretch

INTERVENTIONS:
Other: Passive static stretch — Each experimental group will be submitted to 10 (ten) sessions, with three (3) weekly sessions of static passive stretching, with a 48 h interval between them. Each session will be performed 3 (three) maneuvers containing a duration of 30 seconds, this being the same rest time, performed in all experimental groups.
  Arms: Experimental Group 1; Experimental Group 2; Experimental Group 3

SUMMARY:
Intensity is a "qualitative" variable of a muscle stretching protocol, which is very little studied due to its inherent characteristic of the individual being stretched. However, it was pointed out as an important factor for ADM gain. To verify the effects of different intensities of static passive stretching on flexibility, neuromuscular and functional performance in soccer athletes.

DETAILED DESCRIPTION:
It is a randomized, controlled, clinical trial, composed of male subjects, soccer players, randomly divided into 4 groups: Control Group (CG), Experimental Group 1 (GE1), Experimental Group 2 (GE2) And Experimental Group 3 (GE3). Initially, the measurements of flexibility (passive and active), neuromuscular (muscular passive torque, electromyographic activity), and functional (vertical jump and shuttle run test) of non-dominant lower limbs, performed before and immediately after the 1st And 48 hours after the last session. The GC will only be submitted for initial evaluation and final re-evaluation. The experimental groups will undergo a protocol of static passive stretching containing 10 sessions, divided into 3 weekly sessions, with 3 maneuvers of 30 s, but with different intensities (Tolerable Maximum Pain, Maximum No Pain Discomfort, and Stretching Sensation Without Discomfort) Established from a PERFLEX-modified visual scale. Groups with higher static passive stretching intensities (Maximum Tolerable Pain and Maximum Painless Discomfort) are expected to have greater gains in flexibility, with no change in muscle passive torque, electromyographic activity and functional performance, while the intensity of Feeling of Stretching without Discomfort (in a comfort zone) provides a greater decrease of the muscular passive torque, without significant change of the flexibility, in individual athletes of soccer. This work may contribute to the clinical practice of health professionals, since it seeks to improve the elaboration of the clinical prescription of protocols of static passive stretching (whether performed by the individual or not), establishing optimal levels of intensity for a given muscle group.

ELIGIBILITY:
Inclusion Criteria:

* (1) being male; (2) age range between 18 and 35 years of age; (3) Body Mass Index (BMI) between 19 and 27; (4) be a soccer player with 4 to 5x weekly training; (5) not participating in lower limb stretching programs; (6) no history of injury, trauma, previous surgeries and lower limb disease in the last 6 months; (7) absence of musculoskeletal, cardiorespiratory and neurological disorders that prevent the accomplishment of evaluation and treatment protocols; (8) not under the action of drugs that cause muscle relaxation or that may inhibit tonic muscle action (9) present a limitation of WMD (muscular shortening degree) with ischiatibial extensibility of less than 165 degrees of active extension of the knee with the hip Flexed at 90 °.

Exclusion Criteria:

* (1) initiate stretching practice involving LLLs in daily activities outside the collection site during the study period; (2) not performing any of the evaluation and / or intervention procedures; (3) discontinuance in participating in the research.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-05-09 (Actual); Primary Completion 2017-09-30 (Estimated); Study Completion 2017-11-30 (Estimated)

PRIMARY OUTCOMES:
Range of motion (ROM) | 48 h after intervention
  The measurement will be performed in two positions: with hip flexed at 90 ° and with extended leg elevation, using goniometry for measurement.

SECONDARY OUTCOMES:
Pleasure after stretching program | 1 minute after intervention
  Each volunteer will be asked shortly after each session what was the pleasure felt in achieving the sensation of stretching, which is indicated by the feeling scale.
Pain after stretching session | 1 minute after intervention
  Measurement from the visual analogue scale of 100 mm.
Functional performance | 48 h after intervention
  Evaluation of functional performance with measures of vertical jump and shuttle run
Electromyographic responses of the hamstring | 48 h after intervention
  Electromyographic responses of the hamstring muscles in performing knee extension and hip flexion
Passive torque | 48 h after intervention
  Isokinetic performance evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Wouber H de Brito Vieira, PhD, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Federal University of Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apostolopoulos N, Metsios GS, Flouris AD, Koutedakis Y, Wyon MA. The relevance of stretch intensity and position-a systematic review. Front Psychol. 2015 Aug 18;6:1128. doi: 10.3389/fpsyg.2015.01128. eCollection 2015. PMID 26347668
- [Background] Behm DG, Bradbury EE, Haynes AT, Hodder JN, Leonard AM, Paddock NR. Flexibility is not Related to Stretch-Induced Deficits in Force or Power. J Sports Sci Med. 2006 Mar 1;5(1):33-42. eCollection 2006. PMID 24198679